CLINICAL TRIAL: NCT02480868
Title: A Prospective Clinical Investigation to Assess Safety and Performance of ARTEBONE as Bone Void Filler in a Single Arthrodesis Procedure of the Ankle (Ankle Joint or Subtalar Joint)
Brief Title: ARTEBONE Bone Void Filler in Arthrodesis Procedure of the Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBS-Bioactive Bone Substitutes Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTEBONE 01
Record Dates: First submitted 2015-04-09; First posted 2015-06-25 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis
Keywords: Primary or secondary osteoarthritis; fusion of the ankle
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARTEBONE (Experimental): Bone Void Filler
  Interventions: Device: ARTEBONE

INTERVENTIONS:
Device: ARTEBONE — 4,3 g Bone Void Filler

SUMMARY:
The purpose of this investigation is to assess safety and performance of ARTEBONE Bone Void Filler in the single arthrodesis procedure.

DETAILED DESCRIPTION:
This is a multi-centre, prospective clinical investigation in subjects in need of a single arthrodesis procedure of the ankle (ankle joint or subtalar joint) to relieve persistent pain due to primary or secondary osteoarthritis.

The objectives of the study are to assess safety and performance of ARTEBONE as Bone Void Filler in the single arthrodesis procedure of the ankle (ankle joint or subtalar joint).

The study will be monitored regularly by Clinical Research Associates (CRAs). Monitoring procedures include one or more visits designed to clarify all prerequisites before the study commences. Interim monitoring visits will take place on a regular basis according to a schedule fixed by mutual agreement. During these visits, the CRA will check for completion of the entries on the Case Report Forms (CRFs), their compliance with the Clinical Investigation Plan (CIP), the standard operating procedures (SOP), Good Clinical Practice and International Organization for Standardization 14155 (ISO 14155), and will compare the CRF entries with the source data, as well as update the Investigator´s File (IF).

Source data verification will be performed in an unassisted way (direct access to source documents), unless otherwise required by the local ethics committee.

The sample size of 30 subjects was considered adequate for the safety and performance evaluation in this indication based on earlier discussions with the authorities.

An interim analyses will be performed for 6 months data. There will be descriptive analysis only and comparison to literature. Literature search has been done according to European Union (EU) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed the independent ethics committee approved informed consent form specific to this investigation prior to enrollment.
2. The patient is diagnosed with primary or secondary osteoarthritis requiring fusion of the ankle joint (tibiotalar) or the subtalar joint.
3. The fusion site should be able to be rigidly stabilized with two or three screws across the fusion site.
4. The patient is independent, ambulatory, and could comply with all post-operative evaluations and visits.
5. The patient is at least 18 years of age and considered to be skeletally mature.

Exclusion Criteria:

1. The patient has undergone previous fusion surgery of the proposed fusion site.
2. The fusion site requires other than screw fixation, more than three screws across the fusion site to achieve rigid fixation, or more than one kit (3 cc) of graft material.
3. There is radiographic evidence of bone cysts, segmental defects or growth plate fracture around the fusion site that may negatively impact bony fusion.
4. The patient currently has untreated malignant neoplasm(s) at the surgical site, or is currently undergoing radio- or chemotherapy.
5. The patient has severe diabetes with neuropathy.
6. The patient has a metabolic disorder known to adversely affect the skeleton, other than primary osteoporosis or diabetes (e.g., renal osteodystrophy or hypercalcemia).
7. The patient uses chronic medications known to affect the skeleton (e.g., glucocorticoid usage > 10 mg/day).
8. The patient uses immunosuppressive treatment or medication for osteoporosis.
9. The patient has systemic or severe local inflammation or infections.
10. The patient has a pre-fracture neuromuscular or musculoskeletal deficiency which might limit the ability to perform objective functional measurements.
11. The patient is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.) to the extent that the investigator judges the patient to be unable or unlikely to remain compliant.
12. The patient has an allergy to reindeer protein.
13. The patient has received an investigational therapy or approved therapy for investigational use within 30 days of surgery.
14. The patient is a prisoner, known or suspected to be transient, or has a history of drug/alcohol abuse within the 12 months prior to screening for study entry.
15. The patient is pregnant or a female intending to become pregnant during the study period.
16. The patient is deemed morbidly obese (body mass index [BMI] > 45 kg/m2).
17. The patient has a recent history of smoking during the past six months prior to screening for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
The incidence of unanticipated serious adverse device effects | Before or at 12 months
Bone fusion rates | At 6 months (plus or minus 2 weeks)
  Bone fusion rates assessed by sequential post-operative radiographs and Computer tomography at 6 months (both evaluated by two independent radiologists).
Bone fusion rates | At 12 months (plus or minus 2 weeks)
  Bone fusion rates assessed by sequential post-operative radiographs at 12 months (evaluated by two independent radiologists).

SECONDARY OUTCOMES:
Adverse events | Within 12 months
  Adverse events recorded either voluntarily by the subject in response to a non-leading question (i.e. "how have you been feeling?") or following a clinical observation.
  All adverse events will be assessed by the investigator according to their severity, relationship to the investigational product, action taken, and outcome status as defined in the ISO14155 guideline.
Time-points for returning to work | Within 12 months
  Secondary performance endpoint
Functional performance (Scores of American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale) | 6 months (plus or minus 2 weeks)
  Functional performance at 6 months, secondary performance endpoint
Functional performance (Scores of American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale) | 12 months (plus or minus 2 weeks)
  Functional performance at 12 months, secondary performance endpoint
Subjective pain evaluation (VAS) for fusion site and at weight bearing | 12 weeks (plus or minus 1 week)
  Secondary performance endpoint
Subjective pain evaluation (VAS) for fusion site and at weight bearing | 6 months (plus or minus 2 weeks)
  Secondary performance endpoint
Subjective pain evaluation (VAS) for fusion site and at weight bearing | 12 months (plus or minus 2 weeks)
  Secondary performance endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Juhana Leppilahti, Professor, Principal Investigator — Oulu University Hospital
Locations (5):
- Finland (4):
  - Central Hospital of Central Finland, Jyväskylä
  - South Karelia Central Hospital, Lappeenranta
  - Oulu University Hospital, Oulu
  - Helsinki University Central Hospital Peijas, Vantaa
- Autonomous Public Clinical Hospital No. 1 of Pomeranian Medical University in Szczecin named after professor Tadeusz Sokołowski, Szczecin, Poland